CLINICAL TRIAL: NCT05192148
Title: Seroprevalence of Antibodies to Surface Antigens and Toxins of Clostridioides Difficile
Acronym: PREVADIFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PREVADIFF
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): On the day of inclusion, as part of the research, an additional blood sample will be taken (2 dry tubes of 7 ml each).
  Interventions: Other: Patients

INTERVENTIONS:
Other: Patients — On the day of inclusion, as part of the research, an additional blood sample will be taken (2 dry tubes of 7 ml each).

SUMMARY:
Data on the seroprevalence of antibodies to Clostridioides difficile surface proteins and toxins are scarce.

In 1983, Viscidi et al. showed that antibodies to C. difficile toxins A and B were detected in 60 to 70% of an adult population. Two-thirds of the adults tested had a serological trace, probably linked to a previous encounter with C. difficile.

One of the hypotheses raised would be that exposure to this pathogen occurs very early and regularly throughout our lives. Indeed, in this study, antibodies to C. difficile toxins were detected from early childhood and persisted over time even after 60 years. The antibody response did not appear to vary with age or terrain. However, these results were only qualitative and did not allow for inter-individual variations due to the limitations of the techniques used at the time. Finally, in this work, it was important to underline that the neutralizing character of the cytotoxic effect of toxins on cell culture was not observed in all patients.

Since this seminal work, several studies have shown that the host immune response plays a central role in the pathophysiology of C. difficile infections (CDI). In 2000, Kyne et al. showed that after colonization with a toxigenic C. difficile strain, patients with asymptomatic carriage had significantly higher serum levels of IgG directed against toxin A than patients who developed disease. Subsequently, they also showed in 2001 that a serum response directed against toxin A after a first episode of CDI was associated with less recurrence. Finally, Leav et al. showed in 2010 that a serum response directed against C. difficile toxin B was also associated with protection against recurrent forms.

Several studies have also suggested that the host immune response, this time directed against colonization factors, could also play a major role in the evolution and prognosis of CDI. In a previous study, investigators showed a significant difference in the level of anti-SlpA antibodies (S-layer component) between CDI patients and control patients.

At the same time, the epidemiology of CDI has changed since 2003 due to the emergence of a new epidemic and hypervirulent strain (PCR ribotype 027) producing a third toxin, the binary toxin. The humoral response to this toxin remains poorly described to date.

On the basis of these numerous studies, new therapeutic immunization strategies (active or passive) aimed at neutralizing the action of C. difficile toxins and colonization factors have been or are being developed.

However, it remains to identify the patients likely to benefit from these innovative strategies. This was the main objective of the SERODIFF study (currently being finalized), which identified certain patient profiles in which no seroconversion or isotype class switching of antibodies was observed following CDI. The absence of neutralizing antibody production would seem to correlate with recurrent forms. Thus, these patients would be those who could be eligible for a passive immunization strategy such as the administration of anti-toxin B monoclonal antibodies, bezlotoxumab, recently marketed in France.

In this study, investigators aim to evaluate the seroprevalence stratified by age group, sex and by the main risk factors for CDI. Furthermore, the neutralizing and protective effect of the detected antibodies against C. difficile virulence factors will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years) hospitalized in targeted short-stay (MCO) and long-stay (LTC) services for each of the three identified regions
* French-speaking patient
* Patient affiliated to the social security system or, failing that, to another health insurance system
* Patient able to give free, informed and written consent

Exclusion Criteria:

* History of blood transfusion, vascular filling, dialysis or polyvalent immunoglobulin infusion.
* Patient deprived of liberty
* Patient under court protection
* Patient in an emergency situation
* Patients unable to give personal consent, including adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall seroprevalence of antibodies to the major virulence factors of Clostridioides difficile | Day 1
  This outcome corresponds to the percentage of patients with antibodies detected against each of the antigens studied (toxins and Clostridioides difficile colonization factors).

SECONDARY OUTCOMES:
Immune response profiles | Day 1
  This outcome corresponds to the comparison of antibody positivity rates according to different groups such as gender, age groups, geographical location and community or hospital status.
Observed immune responses | Day 1
  This outcome corresponds to the distribution of serum antibody titers to each antigen of interest (IgG and IgM) and rate of patients with neutralizing antibodies (cell culture cytotoxicity test) among patients with detectable antibodies.
Determination of the seroprevalence of antibodies directed specifically against binary toxins | Day 1
  This outcome corresponds to the percentage of patients with antibodies to C. difficile binary toxins.

CONTACTS AND LOCATIONS:
Overall Officials: Alban LE MONNIER, MD, PhD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (5):
- France (5):
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Hôpital Sainte-Marie Paris, Paris
  - Centre de SSR Pierre Chevalier, Toulon
  - Hôpital d'Instruction des Armées Sainte Anne,, Toulon
  - Centre Hospitalier de Valenciennes, Valenciennes

REFERENCES:
- [Background] Viscidi R, Laughon BE, Yolken R, Bo-Linn P, Moench T, Ryder RW, Bartlett JG. Serum antibody response to toxins A and B of Clostridium difficile. J Infect Dis. 1983 Jul;148(1):93-100. doi: 10.1093/infdis/148.1.93. PMID 6886489
- [Background] Rousseau C, Poilane I, De Pontual L, Maherault AC, Le Monnier A, Collignon A. Clostridium difficile carriage in healthy infants in the community: a potential reservoir for pathogenic strains. Clin Infect Dis. 2012 Nov;55(9):1209-15. doi: 10.1093/cid/cis637. Epub 2012 Jul 25. PMID 22843784
- [Background] Kyne L, Warny M, Qamar A, Kelly CP. Asymptomatic carriage of Clostridium difficile and serum levels of IgG antibody against toxin A. N Engl J Med. 2000 Feb 10;342(6):390-7. doi: 10.1056/NEJM200002103420604. PMID 10666429
- [Background] Kyne L, Warny M, Qamar A, Kelly CP. Association between antibody response to toxin A and protection against recurrent Clostridium difficile diarrhoea. Lancet. 2001 Jan 20;357(9251):189-93. doi: 10.1016/S0140-6736(00)03592-3. PMID 11213096
- [Background] Leav BA, Blair B, Leney M, Knauber M, Reilly C, Lowy I, Gerding DN, Kelly CP, Katchar K, Baxter R, Ambrosino D, Molrine D. Serum anti-toxin B antibody correlates with protection from recurrent Clostridium difficile infection (CDI). Vaccine. 2010 Jan 22;28(4):965-9. doi: 10.1016/j.vaccine.2009.10.144. Epub 2009 Nov 24. PMID 19941990
- [Background] Aboudola S, Kotloff KL, Kyne L, Warny M, Kelly EC, Sougioultzis S, Giannasca PJ, Monath TP, Kelly CP. Clostridium difficile vaccine and serum immunoglobulin G antibody response to toxin A. Infect Immun. 2003 Mar;71(3):1608-10. doi: 10.1128/IAI.71.3.1608-1610.2003. PMID 12595488
- [Background] Lowy I, Molrine DC, Leav BA, Blair BM, Baxter R, Gerding DN, Nichol G, Thomas WD Jr, Leney M, Sloan S, Hay CA, Ambrosino DM. Treatment with monoclonal antibodies against Clostridium difficile toxins. N Engl J Med. 2010 Jan 21;362(3):197-205. doi: 10.1056/NEJMoa0907635. PMID 20089970
- [Background] Gerding DN, Kelly CP, Rahav G, Lee C, Dubberke ER, Kumar PN, Yacyshyn B, Kao D, Eves K, Ellison MC, Hanson ME, Guris D, Dorr MB. Bezlotoxumab for Prevention of Recurrent Clostridium difficile Infection in Patients at Increased Risk for Recurrence. Clin Infect Dis. 2018 Aug 16;67(5):649-656. doi: 10.1093/cid/ciy171. PMID 29538686